CLINICAL TRIAL: NCT04128761
Title: Reinforcer Pathology 1B: Decreasing the Temporal Window
Brief Title: Decreasing the Temporal Window in Individuals With Alcohol Use Disorder
Acronym: RP1B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); McMaster University (Other); Arizona State University (Other); Carilion Clinic (Other); University of Kentucky (Other)
Responsible Party: Principal Investigator, Stephen LaConte, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: #23-621; R01AA027381-01A1 (NIH)
Record Dates: First submitted 2019-10-10; First posted 2019-10-16 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder
Keywords: Delay Discounting; Behavioral Economic Demand; Scarcity Narrative; Alcohol Craving
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scarcity Narrative (Experimental): Participants assigned to the scarcity group will be asked to listen and consider a hypothetical narrative about a sudden loss of resources.
  Interventions: Behavioral: Scarcity Narrative
- Neutral Narrative (Sham Comparator): Participants assigned to the neutral group will be asked to listen and consider a hypothetical narrative about a neutral change in resources.
  Interventions: Behavioral: Neutral Narrative

INTERVENTIONS:
Behavioral: Scarcity Narrative — Participants are presented with a hypothetical scarcity narrative and asked to listen and consider the scenario.
  Arms: Scarcity Narrative
Behavioral: Neutral Narrative — Participants are presented with a hypothetical neutral narrative and asked to listen and consider the scenario.
  Arms: Neutral Narrative

SUMMARY:
In the absence of sufficient monetary resources, individuals must attend to immediate, minimum needs (e.g., food, shelter). This constricts one's temporal window and engenders neglect of the future. In observational studies, scarcity is associated with higher rates of delay discounting. Additionally, socioeconomic status is inversely associated with alcohol use disorder and related problems. Experimentally, scarcity shortens attention, impedes cognitive function, and increases delay discounting in multiple populations. Moreover, scarcity increases demand for fast foods in the obese and increases craving for alcohol in problem drinkers. These data suggest that economic scarcity worsens both components of reinforcer pathology (delay discounting and alcohol overvaluation), thus increasing vulnerability to alcohol use disorder. However, studies investigating the effects of scarcity on alcohol demand discounting rate have been limited. The purpose of Aim 1b is to examine effects of decreasing the temporal window and its concomitant effects on alcohol valuation (demand, and craving) and delay discounting.

DETAILED DESCRIPTION:
Participants will be randomly assigned to experimental or control groups, balanced by discounting rates and sex. We plan to have 112 participants complete the study, based on our power analysis. Participants will complete two online sessions. During the first session, they will complete the baseline assessments. During the second session, they will complete the same assessments after being exposed to the scarcity or control narratives (both in audio format).

The assessment will include delay discounting and demand tasks, and measures of alcohol craving. Participants will also complete assessments of their stress and mood response to the narrative intervention, using the Stress Appraisal Measure (SAM) for two purposes. That is, 1) to monitor participant safety, 2) to measure the mediating ability of affect on changes in the temporal window.

ELIGIBILITY:
Inclusion Criteria:

* High-risk or harmful drinking (AUDIT>15)
* 21 years of age or older
* Desire to quit or cut down on their drinking, but do not have proximate plans to enroll in treatment for AUD during the study period

Exclusion Criteria:

* having a current unmanaged psychotic disorder
* reporting current pregnancy or lactation
* having dementia

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M LaConte, PhD, Principal Investigator — Fralin Biomedical Research Institute at VTC
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will adhere to all NIH requirements regarding data sharing. Participant data collected in this project will be de-identified and made available on a shared secured data repository. We will also share the analysis results. As part of this process, all investigators will be required to agree to the following conditions: 1) will adhere to the reporting responsibilities; 2) will not redistribute the data beyond the requesting individual and named collaborators; 3) will give appropriate acknowledgement; 4) will not use the data for commercial purposes; and 5) will obtain appropriate ethical approvals.
  Results from research conducted will be shared and disseminated, including: regular project meetings, annual meetings, symposia, workshops, and/or conferences for related groups. Manuscripts will be written and submitted for publication in peer-reviewed journals/conferences, following the NIH Public Access Policy guidelines. All necessary ethical approvals will be obtained.
Time Frame: Data will be made available upon request after dissemination of results.
Access Criteria: Data requests will be reviewed by the principal investigator and data will be shared with the expectation of acknowledgment of funding source and primary study team.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Scarcity Narrative | Neutral Narrative
Started | 62 | 62
Completed | 57 | 56
Not Completed | 5 | 6
Not completed — Lost to Follow-up | 5 | 6

BASELINE CHARACTERISTICS:
Population: A total of 124 participants enrolled in the study, with 112 participants (the proposed sample size) completing both sessions. We had additional attrition in the data inspection stage. Participants were included in the analyses if they: 1) completed both sessions, and 2) passed all attention checks programmed in the surveys for both sessions.
Groups:
- Total: Total of all reporting groups
Arm/Group | Scarcity Narrative | Neutral Narrative | Total
Number analyzed (Participants) | 40 | 45 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 44 | 83
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.27 (11.22) | 42.84 (10.54) | 42.58 (10.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 27 | 50
  Male | 17 | 18 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 39 | 42 | 81
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 45 | 85

OUTCOME MEASURES:

1. Primary Outcome: Delay Discounting (DD) Rates
Description: DD rates were measured using an adjusting amount task where participants were presented with hypothetical choices between smaller immediate or larger later amounts of money after a range of delays (1 day-25 years). Individual indifference points were calculated for each delay and then used to estimate DD rates for each participant using Mazur's (1987) equation: V = A/(1+kD), where V is the value of the indifference point, A is the amount of the larger delayed reward, k is the discounting rate, and D is the delay. Discounting rates (k) were then natural-logarithmically transformed (ln(k)). Higher ln(k) indicates steeper discounting and greater reward devaluation with increases in delay, while a lower ln(k) reflects shallower discounting and less reward devaluation with increases in delay.
  Changes in ln(k) were compared within-subjects between S1 and S2. Average ln(k) was calculated for each session (S1 and S2) in each condition (scarcity or neutral).
Time Frame: At the first session (S1; baseline measures) and Session 2 (S2; occurs approximately 2-3 days after S1)
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: ln(K-value)
Arm/Group | Scarcity Narrative | Neutral Narrative
Number analyzed (Participants) | 40 | 45
ln(K-value)
  Session 1 | -4.69 (0.38) | -5.15 (0.38)
  Session 2 | -4.92 (0.40) | -5.58 (0.37)
Statistical Analysis 1: Comparison: Scarcity Narrative vs Neutral Narrative; The effects of narrative type on delay discounting rates were evaluated using a two-way (Scarcity vs. Session) repeated-measures ANOVA; Test type: Other — Mechanistic study examining the influence of scarcity narratives on delay discounting; p = .60, ANOVA — The reported p-value is for the Scarcity and Session interaction

2. Primary Outcome: Intensity of Alcohol Demand
Description: Participants completed a hypothetical Alcohol Purchase Task where they had to indicate how many drinks they would purchase at different prices ($0 to $80 per drink). The number of drinks purchased at $0 was used to calculate the intensity of demand. Changes in intensity of alcohol demand were compared within-subjects between Session 1 and Session 2, and between narrative type (scarcity or neutral).
Time Frame: At the first session (S1; baseline measures) and Session 2 (S2; occurs approximately 2-3 days after S1)
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: Drinks
Arm/Group | Scarcity Narrative | Neutral Narrative
Number analyzed (Participants) | 40 | 45
Drinks
  Session 1 | 14.17 (1.53) | 16.22 (2.55)
  Session 2 | 11.95 (1.26) | 14.91 (2.37)
Statistical Analysis 1: Comparison: Scarcity Narrative vs Neutral Narrative; The effects of narrative type on intensity of alcohol demand were evaluated using a two-way (Scarcity vs. Session) repeated-measures ANOVA; Test type: Other — Mechanistic study examining the influence of scarcity narratives on intensity of demand (i.e., consumption at $0); p = .54, ANOVA — The p-value reported is for the Scarcity and Session interaction term of the two-way repeated-measures ANOVA

3. Primary Outcome: Change in Alcohol Craving
Description: A brief questionnaire (the Alcohol Urges Questionnaire) will be used to assess alcohol craving. The Alcohol Urges Questionnaire is an 8-item survey that produces scores between 8-56, where higher scores indicate greater craving. Change in alcohol craving will be compared within-subjects between Session 1 and Session 2. The scores will be compared between groups (arms) across sessions.
Time Frame: At the first session (S1; baseline measures) and Session 2 (S2; occurs approximately 2-3 days after S1)
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Scarcity Narrative | Neutral Narrative
Number analyzed (Participants) | 40 | 45
score on a scale
  Session 1 | 34.4 (1.98) | 33.11 (1.87)
  Session 2 | 32.17 (2.23) | 32.58 (1.83)
Statistical Analysis 1: Comparison: Scarcity Narrative vs Neutral Narrative; The effects of narrative type alcohol craving were evaluated using a two-way (Scarcity vs. Session) repeated-measures ANOVA; Test type: Other — Mechanistic study examining the influence of scarcity narratives on alcohol craving; p = .88, ANOVA — The p-value reported is for the Scarcity and Session interaction term of the two-way repeated-measures ANOVA

4. Secondary Outcome: Change in Stress Appraisal Measure
Description: The Stress Appraisal Measure will be used to measure acute stress induced by the intervention. This measure is a 28-item survey that produces scores between 28-140, where higher scores indicate greater stress. Change scores were compared between groups during Session 2, to assess differences in stress level as a function of the narrative presented.
Time Frame: Session 2 (occurs approximately 2-3 days after baseline [S1])
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Scarcity Narrative | Neutral Narrative
Number analyzed (Participants) | 40 | 45
score on a scale | 88.52 (2.14) | 73.49 (2.02)
Statistical Analysis 1: Comparison: Scarcity Narrative vs Neutral Narrative; The effects of narrative type on stress was evaluated using a one-way ANOVA; Test type: Other — Mechanistic study examining the influence of scarcity narratives on stress; p < .001, ANOVA

ADVERSE EVENTS:
Time Frame: During study participation (approximately 1 week)
Description: These procedures are not more than minimal risk.
Arm/Group | Scarcity Narrative | Neutral Narrative
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 0/62 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/61/NCT04128761/Prot_SAP_000.pdf